CLINICAL TRIAL: NCT02680197
Title: Randomised, Double Blind, Placebo-controlled, Incomplete Block, 3-way Cross-over Study to Evaluate Efficacy and Safety of 4 Doses of Glycopyrronium Bromide (CHF5259) DPI in Moderate to Severe Patients With COPD
Brief Title: Study to Evaluate Efficacy/Safety of 4 Doses of CHF5259 Via Dry Powder Inhaler (DPI) in Patients With COPD
Acronym: GlycoNEXT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-06302AA1-01; 2015-000558-40 (EudraCT Number)
Record Dates: First submitted 2016-02-04; First posted 2016-02-11 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CHF5259 12.5 μg total daily dose (Experimental): CHF5259 or Placebo administration:
  Patient receives during 4 weeks (28 days) the following treatment : 1 puff of CHF5259 DPI 6.25μg + 1 puff of CHF5259 DPI matched placebo twice a day
  Day 1 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Day 14: pre-dose spirometry
  Day 28 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Interventions: Drug: CHF5259 or Placebo administration
- CHF5259 25 μg total daily dose (Experimental): CHF5259 or Placebo administration: Patient receives during 4 weeks (28 days) the following treatment : 1 puff of CHF5259 DPI 6.25μg + 1 puff of CHF5259 DPI 6.25μg twice a day
  Day 1 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Day 14: pre-dose spirometry
  Day 28 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Interventions: Drug: CHF5259 or Placebo administration
- CHF5259 50 μg total daily dose (Experimental): CHF5259 or Placebo administration: Patient receives during 4 weeks (28 days) the following treatment : 1 puff of CHF5259 DPI 12.5 μg + 1 puff of CHF5259 DPI 12.5 μg twice a day
  Day 1 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Day 14: pre-dose spirometry
  Day 28 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Interventions: Drug: CHF5259 or Placebo administration
- CHF5259 100μg total daily dose (Experimental): CHF5259 or Placebo administration: Patient receives during 4 weeks (28 days) the following treatment :1 puff of CHF5259 DPI 25 μg + 1 puff of CHF5259 DPI 25 μg twice a day
  Interventions :
  Day 1 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Day 14: pre-dose spirometry
  Day 28 : pre-dose spirometry, serial spirometry, Haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Interventions: Drug: CHF5259 or Placebo administration
- CHF5259 matched Placebo BID (Placebo Comparator): CHF5259 or Placebo administration: Patient receives during 4 weeks (28 days) the following treatment : 2 puffs of CHF5259 DPI matched placebo twice a day
  Interventions :
  Day 1 : pre-dose spirometry, serial spirometry, haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Day 14: pre-dose spirometry
  Day 28 : pre-dose spirometry, serial spirometry, haematology/chemistry sample and analyses, BDI/TDI (Baseline and transition dyspnea Indexes), Electrocardiogram
  Interventions: Drug: CHF5259 or Placebo administration

INTERVENTIONS:
Drug: CHF5259 or Placebo administration — Administration of 2 puffs of treatment in the morning and in the evening during a 4 week period. Each patient will be allocated to 3 out of the 5 possible treatments.

SUMMARY:
The study was designed to investigate the efficacy and safety of different doses CHF5259 a long acting muscarinic antagonist in patients with moderate to severe COPD.

DETAILED DESCRIPTION:
Outpatients attending the hospital clinics/study centres will be recruited. Patients with moderate to severe COPD airflow obstruction according to GOLD 2015 criteria.

A total of approximately 300 patients will be enrolled.

Patients are followed during 3 different treatment periods of 4 weeks separated each by 3 weeks wash-out period. The study lasts approximately 21 weeks for each patient and a total of 11 clinic visits is performed during the study.

The primary endpoint is the Forced Expiratory Volume in 1 second (FEV1) Area Under the Curve (AUC) 0-12h normalised by time on Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 40 years
2. Patients with a diagnosis of stable COPD at least 12 months before screening visit.
3. Current smoker or ex-smoker with a smoking history of at least 10 pack-years
4. - A post-bronchodilator FEV1 ≥ 40% and ≤70% of the predicted normal value and,

   * a post-bronchodilator FEV1/FVC < 0.7 and,
   * a change in FEV1 from the pre-bronchodilator value (reversibility) of at least 5% at screening
5. Patients under bronchodilators with long-acting muscarinic antagonist or long-acting 2 agonist (monotherapy or dual therapy), or patients under ICS + LABA (long-acting beta2-agonist) or ICS (Inhaled Corticosteroids) + LAMA (Long Acting Muscarinic Agonist) for at least 4 weeks prior to screening.

   (Patients with a FEV1<50% of the predicted value and a history of 1 exacerbation within the last 12 months must have been treated with ICS+LABA or ICS+LAMA before screening)
6. Ability and cooperative attitude to understand and to perform required outcome measurements of the protocol (e.g. spirometry manoeuvres) and ability to understand the risks involved. Ability to be trained to use the dry powder inhalers.

Exclusion Criteria:

1. Diagnosis of asthma or other respiratory disorders (other than COPD) which may interfere with data interpretation according to the investigator's opinion.
2. Patients had a COPD exacerbation or a lower respiratory tract infection within 8 weeks prior to screening, or during the run-in period, that resulted in the use of an antibiotic, or oral or parenteral corticosteroids, or hospitalisation.
3. Patients with a history of ≥ 2 exacerbations within the last 12 months prior to screening.
4. Patients treated with oral/parenteral β2-agonists or nebulised bronchodilators or phosphodiesterase inhibitors or who received LABA/LAMA/ICS treatment therapy in the 4 weeks prior to screening and during the run-in period.
5. Patient is on an inhaled corticosteroid that has been initiated, or the effective dose has been changed, within 4 weeks prior to screening or during the run-in period (patients on stable dose of ICS for at least 4 weeks prior to screening are allowed).
6. Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia.
7. Patients with known respiratory disorders other than COPD including but not limited to alpha1 antitrypsin deficiency, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension and interstitial lung disease.
8. Patients with medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic.
9. Patients who have unstable concurrent disease that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study;
10. Patients who have a concomitant disease of poor prognosis (e.g., cancer...).
11. Patients who have clinically significant cardiovascular condition diagnosed in the last 6 months
12. Patients with known atrial fibrillation (AF):

    1. Paroxysmal Atrial Fibrillation
    2. Persistent
    3. Long standing persistent.
    4. Permanent
13. Patients with a clinically significant abnormal 12-lead ECG that might, in the judgment of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study.
14. Patients whose electrocardiogram 12-lead ECG shows a QTcF>450 ms for males or QTcF > 470 ms for females.
15. Patients with clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study.
16. Pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS they are willing to use a highly effective birth control methods
17. Patients known to have intolerance/hypersensitivity or any contra-indication to treatment with M3 Antagonist or any of the excipients contained in the formulations used in the study.
18. Patients who have evidence of alcohol or drug abuse, not compliant with the study protocol or not compliant with the study treatments according to investigator's judgment.
19. Patients with major surgery in the previous 3 months or planned during the trial which may affect patient's compliance in study procedures.
20. Patients who have participated in another clinical trial with an investigational drug in the 2 months preceding the screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
FEV1 AUC0-12h normalised by time (L) | Day 28

SECONDARY OUTCOMES:
Change from baseline in morning pre-dose FEV1 (L) | Day 28
Change from baseline in morning pre-dose FEV1 (L) | Day 14
Peak0-4h effect in FEV1 (L) | Day 28
Adverse events and adverse drug reactions | Day 28
Change from baseline in morning pre-dose Forced Vital Capacity FVC (L) | Day 28
Change from baseline in morning pre-dose FVC (L) | Day 14
Change from baseline in morning pre-dose Inspiratory Capacity IC (L) | Day 28
Change from baseline in morning pre-dose IC (L) | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Michael BEEH, MD, Principal Investigator — Institut fuer Atemwegsforschung GmbH
Locations (30):
- Czechia (7):
  - Clinical Trial Site 203-002, Karlovy Vary
  - Clinical Trial Site 203-003, Kralupy nad Vltavou
  - Clinical Trial Site 203-001, Mělník
  - Clinical Trial Site 203-007, Mladá Boleslav
  - Clinical Trial Site 203-005, Moravský Krumlov
  - Clinical Trial Site 203-006, Teplice
  - Clinical Trial Site 203-004, Varnsdorf
- Germany (6):
  - Clinical Trial Site 276-003, Bonn
  - Clinical Trial Site 276-004, Cottbus
  - Clinical Trial Site 276-006, Freiburg im Breisgau
  - Clinical Trial Site 276-002, Großhansdorf
  - Clinical Trial Site 276-005, Stuttgart
  - Clinical Trial Site 276-001, Wiesbaden
- Hungary (9):
  - Clinical Trail Site 348-006, Budapest
  - Clinical Trial Site 348-003, Budapest
  - Clinical Trial Site 348-004, Budapest
  - Clinical Trial Site 348-001, Deszk
  - Clinical Trial Site 348-005, Komárom
  - Clinical Trial Site 348-002, Létavértes
  - Clinical Trail Site 348-008, Miskolc
  - Clinical Trail Site 348-009, Seregélyes
  - Clinical Trail Site 348-007, Szombathely
- Romania (8):
  - Clinical Trial Site 642-005, Bacau
  - Clinical Trial Site 642-003, Brasov
  - Clinical Trial Site 642-007, Bucharest
  - Clinical Trial Site 642-008, Bucharest
  - Clinical Trial Site 642-004, Cluj-Napoca
  - Clinical Trial Site 642-001, Codlea
  - Clinical Trial Site 642-002, Miercurea-Ciuc
  - Clinical Trial Site 642-006, Suceava

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beeh KM, Emirova A, Prunier H, Santoro D, Nandeuil MA. Dose-response of an extrafine dry powder inhaler formulation of glycopyrronium bromide: randomized, double-blind, placebo-controlled, dose-ranging study (GlycoNEXT). Int J Chron Obstruct Pulmon Dis. 2018 May 25;13:1701-1711. doi: 10.2147/COPD.S168493. eCollection 2018. PMID 29872288
- See also: Study Record on EU Clinical Trials Register including results — http://www.clinicaltrialsregister.eu/ctr-search/trial/2015-000558-40/results